CLINICAL TRIAL: NCT06615622
Title: A Comparative Study of Peripheral Nerve Ultrasound Findings in Immune Mediated Peripheral Nerve Disorders; a Hospital-based Study
Brief Title: Our Study Aims to Determine if Nerve Alterations in Acute GBS and CIDP Detectable by Ultrasound Match Electrodiagnostic Findings and if This Method Aids Early Diagnosis, Predict Their Outcomes and Differentiate Between Axonal and Demyelinating Subtypes.
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Gad Ibrahim Farghly, Principal Investigator, Assiut University
Other Study IDs: 04-2024-200877
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Guillain Barré Syndrome; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Peripheral Nerve Disorder; Peripheral Nerves US; Peripheral Neuropathy
Keywords: Peripheral nerve ultrasound; immune mediated nerve disorders; Guillain-Barré syndrome; Chronic inflammatory demyelinating polyradiculoneuropathy
MeSH Terms: conditions — Guillain-Barre Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Neuritis; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Serum samples CSF samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Patients with immune mediated peripheral nerve disorders GB syndrome and CIDP
  Interventions: Dietary Supplement: Placebo
- Control: Healthy control matching group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Thiotacid 300 mg tab once/day

SUMMARY:
Neuromuscular ultrasound (NMUS) is emerging as a valuable non-invasive diagnostic tool. In GBS, NMUS can detect proximal nerve enlargement early, before neurophysiological changes. Persistent nerve enlargement can be observed up to 15 years, though its correlation with disability varies. Research is needed to clarify NMUS findings in GBS and CIDP over time. Early detection of nerve root enlargement via NMUS could facilitate earlier diagnosis and intervention, improving patient outcomes and understanding of these conditions' pathophysiology.

This study aims to determine if nerve alterations in acute GBS and CIDP detectable by ultrasound match electrodiagnostic findings and if this method aids early diagnosis. The investigators will perform serial nerve ultrasounds and NCS to investigate nerve morphology, predict outcomes, and differentiate between axonal and demyelinating subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of patient group:

   * GBS Patients: Diagnosed according to the criteria of the National Institute of Neurological Disorders and Stroke (NINDS) and the Brighton Collaboration (2011).
   * CIDP Patients: Diagnosed according to the criteria of the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS).
2. Age: Participants aged 18 to 75 years.
3. Onset:

   * GBS Patients: Recent onset of GBS within the first 2 weeks of symptom onset.
   * CIDP Patients: Either relapsing or progressive course consistent with CIDP diagnosis.
4. Gender: Both male and female participants are eligible.
5. Participation: Willingness to participate in the study, including undergoing disease-related examinations and assessments.
6. Consent: Ability and willingness to provide informed consent

Exclusion Criteria:

1. Patients unable or unwilling to provide informed consent.
2. Patients with metabolic disorders or malignancies.
3. Patients with other causes of peripheral neuropathy.
4. Patients with other causes of acute flaccid paralysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A hospital-based study. Patients who are admitted to Assiut university hospitals, neuropsychiatry department.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Detection of Nerve Alterations via Ultrasound | 6 months
  * Determine if patients with acute GBS and CIDP exhibit nerve alterations detectable by ultrasound that are comparable to electrodiagnostic findings.
  * Assess the utility of ultrasound in diagnosing GBS and CIDP in the very early phase of the disease.

SECONDARY OUTCOMES:
Evaluation of Nerve Morphology Evolution | 6 months
  * Investigate patterns of nerve morphology through nerve ultrasound studies in GBS and CIDP patients over the course of the disease.
  * Compare these patterns with serial NCS findings.
Prediction of Outcomes and Recovery | 6 months
  - Evaluate the potential of nerve ultrasound changes as predictors of clinical outcomes and recovery in GBS and CIDP patients.
Differentiation of Subtypes | 6 months
  - Assess if early nerve ultrasound changes can differentiate between axonal and demyelinating subtypes of GBS and CIDP.
Correlation with Clinical Scales | 6 months
  - Correlate ultrasound findings with clinical scales and outcomes, such as the Guillain-Barré Syndrome Disability Scale (GDS), Medical Research Council Sum Score (MRC sum score), and Erasmus GBS Outcome Scale (EGOS)
Comparison with Healthy Controls | 6 months
  - Compare the ultrasound parameters of GBS and CIDP patients with age and sex-matched healthy controls to identify significant differences in nerve morphology

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hughes RA, Swan AV, Raphael JC, Annane D, van Koningsveld R, van Doorn PA. Immunotherapy for Guillain-Barre syndrome: a systematic review. Brain. 2007 Sep;130(Pt 9):2245-57. doi: 10.1093/brain/awm004. Epub 2007 Mar 2. PMID 17337484
- [Background] Hughes RA, Raphael JC, Swan AV, Doorn PA. Intravenous immunoglobulin for Guillain-Barre syndrome. Cochrane Database Syst Rev. 2004;(1):CD002063. doi: 10.1002/14651858.CD002063.pub2. PMID 14973982
- [Background] Hughes RA, Swan AV, van Doorn PA. Intravenous immunoglobulin for Guillain-Barre syndrome. Cochrane Database Syst Rev. 2014 Sep 19;2014(9):CD002063. doi: 10.1002/14651858.CD002063.pub6. PMID 25238327
- [Background] van den Berg B, Walgaard C, Drenthen J, Fokke C, Jacobs BC, van Doorn PA. Guillain-Barre syndrome: pathogenesis, diagnosis, treatment and prognosis. Nat Rev Neurol. 2014 Aug;10(8):469-82. doi: 10.1038/nrneurol.2014.121. Epub 2014 Jul 15. PMID 25023340
- [Background] Willison HJ, Jacobs BC, van Doorn PA. Guillain-Barre syndrome. Lancet. 2016 Aug 13;388(10045):717-27. doi: 10.1016/S0140-6736(16)00339-1. Epub 2016 Mar 2. PMID 26948435
- [Background] Jacobs BC, Rothbarth PH, van der Meche FG, Herbrink P, Schmitz PI, de Klerk MA, van Doorn PA. The spectrum of antecedent infections in Guillain-Barre syndrome: a case-control study. Neurology. 1998 Oct;51(4):1110-5. doi: 10.1212/wnl.51.4.1110. PMID 9781538
- [Background] Laman JD, Huizinga R, Boons GJ, Jacobs BC. Guillain-Barre syndrome: expanding the concept of molecular mimicry. Trends Immunol. 2022 Apr;43(4):296-308. doi: 10.1016/j.it.2022.02.003. Epub 2022 Mar 4. PMID 35256276
- [Background] Sejvar JJ, Baughman AL, Wise M, Morgan OW. Population incidence of Guillain-Barre syndrome: a systematic review and meta-analysis. Neuroepidemiology. 2011;36(2):123-33. doi: 10.1159/000324710. Epub 2011 Mar 21. PMID 21422765